CLINICAL TRIAL: NCT06922669
Title: Efficacy and Safety of Glucocorticoids for Acute Drug Induced Liver Injury With Hyperbilirubinemia: A Multicenter Randomized Controlled Trial
Brief Title: Glucocorticoids for Acute Drug Induced Liver Injury With Hyperbilirubinemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHNKKY-ASDILI-RCT
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Drug Induced Liver Injury
Keywords: Drug induced liver injury; liver failure; glucocorticoids; clinical trial; Hyperbilirubinemia
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Liver Failure; Hyperbilirubinemia | interventions — Methylprednisolone; 18alpha,20beta-hydroxy-11-oxo-norolean-12-en-3beta-yl-2-O-beta-D-glucopyranurosyl-alpha-D-glucopyranosiduronate magnesium tetrahydrate; Glutathione; Silymarin; polyene phosphatidylcholine; essential 303 forte; Ursodeoxycholic Acid; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoids group (Experimental): Glucocorticoids step-down therapy combined with conventional treatment.
  Interventions: Drug: Methylprednisolone; Drug: Magnesium isoglycyrrhizinate; Drug: Glutathione; Drug: Silymarin; Drug: Polyene Phosphatidylcholine; Drug: Ursodeoxycholic acid capsules; Drug: Ademetionine 1,4-Butanedisulfonate; Procedure: Plaslna exchange; Procedure: Liver transplantation
- Conventional treatment (Active Comparator): Only conventional treatment according to the Chinese practice guidelines regarding the management of DILI.
  Interventions: Drug: Magnesium isoglycyrrhizinate; Drug: Glutathione; Drug: Silymarin; Drug: Polyene Phosphatidylcholine; Drug: Ursodeoxycholic acid capsules; Drug: Ademetionine 1,4-Butanedisulfonate; Procedure: Plaslna exchange; Procedure: Liver transplantation

INTERVENTIONS:
Drug: Methylprednisolone — Initially, an intravenous dose of 1 mg/kg/day of methylprednisolone will be administered for one week, with the possibility of extending treatment to two weeks if necessary. Following this, participants will receive oral methylprednisolone tablets, starting at a dose of 40 mg/day. The oral dosage will be gradually tapered based on the participants' condition over a period of 1 to 3 months.
  Other Names: Medrol
  Arms: Glucocorticoids group
Drug: Magnesium isoglycyrrhizinate — It is suitable for patients with hepatocellular or mixed DILI. A daily dose of 0.15g to 0.2g
Drug: Glutathione — It is suitable for patients with hepatocellular or mixed DILI. A daily dose of 1.2g to 1.8g
Drug: Silymarin — It is suitable for patients with hepatocellular or mixed DILI. The dosage is 140 mg, taken 2 to 3 times per day.
  Other Names: Legalon
Drug: Polyene Phosphatidylcholine — It is suitable for patients with hepatocellular or mixed DILI. The dosage is 228mg-456mg, taken 3 times per day.
  Other Names: Essentiale
Drug: Ursodeoxycholic acid capsules — It is suitable for patients with cholestatic or mixed DILI. A daily dose of 10mg-15mg/kg/day.
  Other Names: Ursofalk
Drug: Ademetionine 1,4-Butanedisulfonate — It is suitable for patients with cholestatic or mixed DILI. A daily dose of 0.5g to 1g.
  Other Names: Transmeti
Procedure: Plaslna exchange — It is suitable for patients whose condition continues to worsen or even develop to liver failure.
  Other Names: Artificial liver support
Procedure: Liver transplantation — It is suitable for patients whose condition continues to worsen or even develop to liver failure.

SUMMARY:
Drug-induced liver injury (DILI) can lead to potentially fatal complications, such as acute liver failure and even death. In clinical practice, glucocorticoids have been considered in some cases of DILI, especially patients with hyperbilirubinemia. However, the available evidence remains controversial and its quality is also very limited. Herein, a multicenter randomized controlled trial (RCT) has been designed to explore the efficacy and safety of glucocorticoids in patients with acute DILI and hyperbilirubinemia.

DETAILED DESCRIPTION:
Overall, 232 patients with acute DILI with hyperbilirubinemia will be enrolled. They will be randomly assigned at a ratio of 1:1 to the conventional treatment alone or combined with glucocorticoids groups. The primary endpoint is the improvement of DILI after treatment on second week. Secondary endpoints include the improvement of DILI on fourth week, rates of progressive liver injury, liver failure, liver transplantation, survival, and adverse events. Exploratory endpoints will assess the beneficial population and changes of inflammatory factors following glucocorticoid treatment.

ELIGIBILITY:
Inclusion Criteria:

* A definite diagnosis of acute DILI;
* 5×ULN ≤ TBIL level at baseline ≤ 20×ULN;
* Age 18-80 years old;
* Sign the informed consent form.

Exclusion Criteria:

* Other causes of liver injury, including viral hepatitis, cytomegalovirus infection, Epstein-Barr virus infection, Herpes virus infection, autoimmune liver disease, alcoholic liver disease, hypoxic/ischemic liver disease, Budd-Chiari syndrome, biliary tract disease, Wilson's disease, hemochromatosis, and α1-antitrypsin deficiency;
* Immune checkpoint inhibitors or gynura segetum induced DILI;
* Absolute contraindications to glucocorticoids, such as systemic mold infections or allergies;
* A history of glucocorticoid therapy within 3 months before enrollment;
* A history of diseases requiring glucocorticoid maintenance therapy, such as rheumatoid arthritis, systemic lupus erythematosus, systemic dermatomyositis, etc;
* A history of liver transplantation;
* Received artificial liver therapy before enrollment;
* Malignant tumor of the liver, bile duct, pancreas or liver metastasis
* Acute liver failure;
* Renal dysfunction, creatinine Cr≥133μmol/L;
* Neutrophil count <1,000,000,000/L;
* Active tuberculosis;
* Severe cardiopulmonary diseases;
* Recent surgery or trauma;
* Mental illness;
* Pregnancy or lactation;
* Participated in other clinical studies within 3 months before enrollment;
* Other conditions judged by the clinician to be inappropriate for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of DILI on the second week | 2 weeks
  TBIL level decreases by 50% as compared to the baseline level.

SECONDARY OUTCOMES:
Improvement of DILI on the fourth week | 4 weeks
  TBIL level decreases by 50% as compared to the baseline level.
Progressive liver injury on the second week | 2 weeks
  TBIL level increases as compared to the baseline level.
Progressive liver injury on the fourth week | 4 weeks
  TBIL level increases as compared to the baseline level.
Improvement of liver enzymes on the second week | 2 weeks
  Proportion of 50% reduction from baseline in ALT, AST, ALP, and GGT levels.
Improvement of liver enzymes on the fourth week | 4 weeks
  Proportion of 50% reduction from baseline in ALT, AST, ALP, and GGT levels.
Liver failure | 3 months
  Participants develop overt hepatic encephalopathy with an INR of ≥1.5.
Liver transplantation | 3 months
  Participants undergo liver transplantation due to liver failure.
Survival | 3 months
  All participants will be followed by telephone to record survival status, including the major cause and date of death.
Adverse events | 3 months
  Adverse events related to glucocorticoids mainly include infection, water-sodium retention, Cushing syndrome, poor glycemic, gastrointestinal ulcer, thromboembolic disease, neuropsychiatric symptoms, osteoporosis, increased intraocular pressure, and withdrawal syndrome. They will be closely recorded during the period of glucocorticoids treatment.

OTHER OUTCOMES:
Population who will be more suitable for glucocorticoids treatment | 3 months
  Characteristics of patients with DILI in whom glucocorticoids treatment is more beneficial.
Changes of inflammatory factors | 4 weeks
  Changes of IL-6 and TNF-α levels.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, Principal Investigator — Department of Gastroenterology, General Hospital of Northern Theater Command; Weifen Xie, Principal Investigator — Shanghai changzheng hospital, Naval Medical University; Xin Zeng, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine; Lu Zhou, Principal Investigator — General Hospital, Tianjin Medical University; Fengmei Wang, Principal Investigator — Tianjin First Central Hospital; Qing Ye, Principal Investigator — Tianjin Third Central Hospital; Yanjing Gao, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hou FQ, Zeng Z, Wang GQ. Hospital admissions for drug-induced liver injury: clinical features, therapy, and outcomes. Cell Biochem Biophys. 2012 Nov;64(2):77-83. doi: 10.1007/s12013-012-9373-y. PMID 22806342
- [Result] Hu PF, Wang PQ, Chen H, Hu XF, Xie QP, Shi J, Lin L, Xie WF. Beneficial effect of corticosteroids for patients with severe drug-induced liver injury. J Dig Dis. 2016 Sep;17(9):618-627. doi: 10.1111/1751-2980.12383. PMID 27426618
- [Result] Chai L, Wang R, Teschke R, Jin S, Deng J, Qi X. Successful corticosteroid therapy for severe liver injury secondary to herbal traditional Chinese medicine, Mega Defends X, assessed for causality by the updated RUCAM: A case report. Medicine (Baltimore). 2024 Aug 23;103(34):e39439. doi: 10.1097/MD.0000000000039439. PMID 39183394
- [Result] Mao Y, Ma S, Liu C, Liu X, Su M, Li D, Li Y, Chen G, Chen J, Chen J, Zhao J, Guo X, Tang J, Zhuge Y, Xie Q, Xie W, Lai R, Cai D, Cai Q, Zhi Y, Li X; Technology Committee on DILI Prevention, Management, Chinese Medical Biotechnology Association; Study Group on Drug-Induced Liver Disease, Chinese Society of Hepatology, Chinese Medical Association. Chinese guideline for the diagnosis and treatment of drug-induced liver injury: an update. Hepatol Int. 2024 Apr;18(2):384-419. doi: 10.1007/s12072-023-10633-7. Epub 2024 Feb 24. PMID 38402364